CLINICAL TRIAL: NCT01975961
Title: A Randomized, Open-label, Single-dose, 2-way Cross-over Study to Compare the Safety and the Pharmacokinetic Characteristics of the Co-administration of Telmisartan and Rosuvastatin and YH16410 in Healthy Volunteers
Brief Title: PK Study of Telmisartan/Rosuvastatin FDC Compared to Combination of Telmisartan and Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: YH16410-102
Record Dates: First submitted 2013-10-20; First posted 2013-11-05 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-10

CONDITIONS: Dyslipidemia & Hypertension
MeSH Terms: conditions — Dyslipidemias; Hypertension | interventions — Rosuvastatin Calcium; Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FDC YH16410 (Experimental): Drug: Test treatment: FDC YH16410 (Telmisartan 80mg/ Rosuvastatin 20mg).
  Subjects will receive single oral dose of 1 tablet of FDC containing Telmisartan 80mg and Rosuvastatin 20mg in fasted state
  Interventions: Drug: Crestor 20mg(Rosuvastatin 20mg), Micardis 80mg(Telmisartan 80mg) , FDC
- Co-administration (Active Comparator): Drug: Reference Treatment: Co-administration(Telmisartan 80mg and Rosuvastatin 20mg).
  Subjects will receive 1 x Telmisartan 80mg with 1 x Rosuvastatin 20mg tablet administered orally in fasted state as a single dose
  Interventions: Drug: Crestor 20mg(Rosuvastatin 20mg), Micardis 80mg(Telmisartan 80mg) , FDC

INTERVENTIONS:
Drug: Crestor 20mg(Rosuvastatin 20mg), Micardis 80mg(Telmisartan 80mg) , FDC — For co-administration, Crestor 1 tablet and Micardis 1 tablet. For FDC administration, FDC 1 tablet.

SUMMARY:
This is a 2 by 2 cross-over study to evaluate pharmacokinetics of telmisartan and rosuvastatin FDC compared to reference telmisartan and rosuvastatin coadministered in two groups enrolling healthy adult male and female subjects under fasting conditions.

Subjects will be admitted to the clinic in the evening before Day 1. All subjects will receive a single oral dose of telmisartan/rosuvastatin FDC or telmisartan and rosuvastatin co-administered in the morning on Day 1. All the subjects will remain in the clinical unit until completion of all assessments on Day 2 including collection post-dose PK sample. Subjects will return to the clinic for pharmacokinetic samples at scheduled time.

The two treatment periods will be separated by a washout period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female aged 20 to 50 with a body mass index(BMI) between 18.5 and 25 kg/m2
2. Acceptable medical history, physical examination, laboratory tests and EKG, during screening
3. Provision of signed written informed consent 20~50 yrs old, healthy Korean Subjects

Exclusion Criteria:

1. History of and clinically significant disease
2. Sitting blood pressure meeting the following criteria at screening: 150 ≥ systolic blood pressure ≤100 (mmHg) and 100 ≥ diastolic blood pressure ≤ 65 (mmHg) amd 100 ≥ Heart rate ≤ 40
3. A history of drug abuse or the presence of positive reactions to drugs that have abuse potential in urine screenings for drugs.
4. Administration of other investigational products within 90 days prior to the first dosing.
5. Administration of herbal medicine within 28 days or administration of ethical drugs within 14 days or administration of over-the-counter (OTC) drugs within 7 days prior to the first dosing of the investigational product (if the investigator (study doctor) determines that the person meets other criteria appropriately, the relevant person may participate in the study).
6. Have AST(SGOT) or/and ALT(SGPT) > 3 times of normal upper limit at the time of screening
7. Volunteers considered not eligible for the clinical trial by the investigator (study doctor) due to reasons including laboratory test results, ECGs, or vital signs.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 185 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
plasma pharmacokinetic parameters for telmisartan and rosuvastatin in relevant treatments | 0~72hr, 17points

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea